CLINICAL TRIAL: NCT05923099
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Multi-site, Parallel-group, Dose-finding Trial to Evaluate the Efficacy and Safety of Different Doses of Subcutaneously Administered LEO 138559 in Adult Subjects With Moderate-to-severe Atopic Dermatitis
Brief Title: A Trial to Evaluate the Efficacy and Safety of Different Doses of LEO 138559 in Adults With Moderate-to-severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP0145-2240; U1111-1286-0955 (Other: World Health Organization (WHO)); 2022-500777-14-00 (EU CTIS Number)
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose regimen 1 (Experimental): Dose A every week from Week 0 to Week 3, then every 2 weeks from Week 4 to Week 16
  Interventions: Drug: LEO 138559
- Dose regimen 2 (Experimental): Dose B every week from Week 0 to Week 2, then every 2 weeks from Week 4 to Week 16
  Interventions: Drug: LEO 138559
- Dose regimen 3 (Experimental): Dose A at Week 0 and Week 2, then dose C every 2 weeks from Week 4 to Week 16
  Interventions: Drug: LEO 138559
- Dose regimen 4 (Experimental): Dose C at Week 0 and Week 2, then dose D every 2 weeks from Week 4 to Week 16
  Interventions: Drug: LEO 138559
- Placebo regimen (Placebo Comparator): Placebo every week from Week 0 to Week 3, then every 2 weeks from Week 4 to Week 16
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LEO 138559 — LEO 138559 given by injection just under the skin
  Other Names: LEO 138559 is also called "temtokibart"
  Arms: Dose regimen 1; Dose regimen 2; Dose regimen 3; Dose regimen 4
Drug: Placebo — Placebo given by injection just under the skin
  Arms: Placebo regimen

SUMMARY:
The purpose of this trial is to test different doses of the trial medicine (LEO 138559) and see how well they work and how safe they are at treating moderate to severe atopic dermatitis in adults. There will be 4 different doses, that will also be compared to a placebo (a dummy medicine that doesn't contain the active ingredient of LEO 138559). Each participant will be randomly assigned to one of the 4 doses of LEO 138559 or placebo. In all arms, injections of placebo may be used to mask the different doses.

The trial will last up to 36 weeks, including a screening/washout period (up to 4 weeks), a treatment period (16 weeks), and a follow up period (16 weeks). The participants will visit the clinic 17 times. For the first 4 weeks of the treatment period, participants will visit the clinic every week. For the next 12 weeks of the treatment period, participants will visit the clinic every 2 weeks. For the 16 week follow up period, participants will visit the clinic every 4 weeks.

The treatments will be given to the participants by staff at the clinic. They are given as an injection just under the skin.

At each visit the doctor will check the participants atopic dermatitis and if they have had any side effects. Participants will also complete an electronic diary every day about their atopic dermatitis and quality of life.

LEO 138559 is also called "Temtokibart".

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent has been obtained prior to any protocol related procedures.
* 18-75 years old (both included) at screening (Visit 1).
* Willingness to comply with the clinical trial protocol.
* At screening, diagnosis of atopic dermatitis (AD) as defined by the Hanifin and Rajka (1980) criteria for AD.

  * History of AD for ≥1 year.
* Subjects who have a recent history (within 12 months before screening) with documented inadequate response to treatment with topical corticosteroid(s) (TCS) (±topical calcineurin inhibitor(s) (TCI) as appropriate) or for whom these topical AD treatments are medically inadvisable (e.g. due to important side effects or safety risks).
* Eczema Area and Severity Index (EASI) score ≥12 at screening and ≥16 at baseline.
* Validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) score ≥3 at screening and baseline.
* Body Surface Area (BSA) of AD involvement ≥10% at screening and baseline.
* Atopic Dermatitis Symptom Diary (ADSD) Worst Itch score (weekly average) ≥4 at baseline.
* A woman of childbearing potential must use a highly effective form of birth control throughout the trial and for at least 18 weeks after last administration of IMP.

Exclusion Criteria:

* Major surgery within 8 weeks prior to screening, or planned inpatient surgery or hospitalization during the trial period.
* Active dermatologic condition that could confound the diagnosis of AD or interfere with assessment of the treatment (e.g. scabies, contact dermatitis, rosacea, urticaria, or psoriasis).
* History of cancer, with the following exceptions:

  * Subjects who have had basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible provided that the subject is in remission and curative therapy was completed at least 12 months prior to screening.
  * Subjects who have had other malignancies are eligible provided that the subject is in remission and curative therapy was completed at least 5 years prior to screening
* History of or current immunodeficiency syndrome.
* History of anaphylaxis following any biologic therapy.
* History of clinically significant infection within 4 weeks prior to baseline which, in the opinion of the investigator, may compromise the safety of the subject in the trial, interfere with evaluation of the IMP, or reduce the subject's ability to participate in the trial.
* Skin infection within 7 days prior to baseline
* Positive HBsAg or positive anti-HCV AND positive HCV RNA at screening.
* History of HIV infection or positive HIV serology at screening.
* Evidence of active or latent tuberculosis according to local standard of care for patients requiring initiation of a biologic treatment.
* ALT or AST level ≥2.0 times the ULN at screening.
* History of attempted suicide or is at significant risk of suicide (either in the opinion of the investigator or defined as a "yes" to suicidal ideation questions no. 4 or 5 or answering "yes" to suicidal behavior on the C-SSRS Screening version).
* Known or suspected hypersensitivity to any component(s) of the IMP.
* Any disorder at screening and/or baseline, which is not stable in the opinion of the investigator, and could:

  * Affect the safety of the subject throughout the trial.
  * Influence the results of the trial.
  * Impede the subject's ability to complete the trial.
* Any significant abnormal finding at screening and/or baseline which may, in the opinion of the investigator:

  * Put the subject at risk because of their participation in the trial.
  * Influence the results of the trial.
  * Influence the subject's ability to complete the trial.
* Current or recent chronic alcohol or drug abuse, or any other condition associated with poor compliance as judged by the investigator.
* Women who are pregnant or breastfeeding.
* Previous treatment with LEO 138559.
* Previous exposure to fezakinumab (anti-IL-22 Ab).
* Systemic treatment with immunosuppressive drugs, immunomodulating drugs, retinoids, corticosteroids (steroid eyedrops and inhaled or intranasal steroids are allowed), or JAK inhibitors within 28 days or 5 half-lives prior to baseline, whichever is longer.
* Use of tanning beds or phototherapy, within 4 weeks prior to baseline.
* Receipt of blood products within 28 days prior to screening.
* Treatment with:

  * Any marketed or investigational biologic agents within 3 months or 5 half-lives, whichever is longer, prior to baseline.
  * Any cell-depleting agents including but not limited to rituximab: within 6 months prior to baseline, or until lymphocyte count returns to normal, whichever is longer.
* Treatment with TCS, TCI, topical PDE-4 inhibitors, topical JAK inhibitors, or other medicated topical treatments within 7 days prior to baseline.
* Receipt of live attenuated vaccines 30 days prior to baseline.
* Treatment with any non-marketed drug substance (that is, an agent which has not yet been made available for clinical use following registration) within the last 4 weeks or 5 half lives prior to randomization, whichever is longer.
* Current participation in any other interventional clinical trial.
* Previously randomized in this clinical trial.
* Employees of the trial site, or any other individuals directly involved with the planning or conduct of the trial, or immediate family members of such individuals.
* Subjects who are legally institutionalized.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-12-11 (Actual); Study Completion 2025-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, Study Director — LEO Pharma
Locations (69):
- United States (12):
  - LEO Investigational Site, Fountain Valley, California
  - LEO Investigational Site, Los Angeles, California
  - LEO Investigational Site, San Francisco, California
  - LEO Investigational Site, Hialeah, Florida
  - LEO investigational site, Indianapolis, Indiana
  - LEO investigational Site, New Albany, Indiana
  - LEO Investigational Site, Ann Arbor, Michigan
  - LEO Investigational Site, New York, New York
  - LEO Investigational Site, Raleigh, North Carolina
  - LEO Investigational Site, Cincinnati, Ohio
  - LEO Investigational Site, Mayfield Heights, Ohio
  - LEO Investigational Site, North Charleston, South Carolina
- Canada (7):
  - LEO Investigational Site, Edmonton, Albana
  - LEO Investigational Site, Calgary, Alberta
  - LEO Investigational Site, Edmonton, Alberta
  - LEO Investigational Site, Surrey, British Columbia
  - LEO Investigational Site, Mississauga, Ontario
  - LEO Investigational Site, Sherbrooke, Quebec
  - LEO Investigational Site, Verdun, Quebec
- Czechia (3):
  - LEO Investigational Site, Náchod
  - LEO Investigatonal Site, Ostrava-Poruba
  - LEO Investigational Site, Prague
- France (5):
  - LEO Investigational Site, Martigues, Bouches-du-Rhône
  - LEO Investigational Site, Dijon
  - LEO Investigational Site, Nice
  - LEO Investigational Site, Paris
  - LEO Investigational Site, Rouen
- Germany (11):
  - LEO Investigational Site, Augsburg
  - LEO Investigational Site, Bad Bentheim
  - LEO Investigational Site, Berlin
  - LEO Investigational Site, Dresden
  - LEO Investigational Site, Frankfurt am Main
  - LEO Investigational Site, Freiburg im Breisgau
  - LEO Investigational Site, Gera
  - LEO Investigational Site, Kiel
  - LEO Investigational Site, Leipzig
  - LEO Investigational Site, Mahlow
  - LEO Investigational Site, Münster
- Hungary (3):
  - LEO Investigational Site, Debrecen
  - LEO Investigational Site, Pécs
  - LEO Investigational Site, Szeged
- Japan (7):
  - LEO Investigational Site, Fukuoka, Fukuoka
  - LEO Investigational Site, Kobe, Hyōgo
  - LEO Investigational Site, Yokohama, Kanagawa
  - LEO Investigational Site, Takatsuki-shi, Osaka
  - LEO Investigational Site, Koto-ku, Tokyo
  - LEO Investigational Site, Takaoka-shi, Toyama
  - LEO Investigational Site, Tokyo
- Poland (5):
  - LEO Investigational Site, Wroclaw, Lower Silesian Voivodeship
  - LEO Investigational Site, Krakow
  - LEO Investigational Site, Malbork
  - LEO Investigational Site, Mikołów
  - LEO Investigational Site, Wroclaw
- Romania (3):
  - LEO Investigational Site, Cluj-Napoca
  - LEO Investigational Site, Iași
  - LEO Investigational Site, Timișoara
- Spain (7):
  - LEO Investigational Site, Badalona, Barcelona
  - LEO Investigational Site, Alcobendas
  - LEO Investigational Site, Alicante
  - LEO Investigational Site, Barcelona
  - LEO Investigational Site, Córdoba
  - LEO Investigational Site, Madrid
  - LEO Investigational Site, Zaragoza
- United Kingdom (6):
  - LEO Investigational Site, Edinburgh
  - LEO Investigational Site, Harrow
  - LEO Investigational Site, London
  - LEO Investigational Site, Manchester
  - LEO Investigational Site, Southampton
  - LEO Investigational Site, Walsall

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at sites in 11 countries (Canada, Czech Republic, France, Germany, Hungary, Japan, Poland, Romania, Spain, United Kingdom, and United States).
Pre-assignment Details: Participants were randomized 1:1:1:1:1 to 5 different treatment groups (4 different dose regimens of LEO 138559 and placebo).
Groups:
- Dose Regimen 1: Dose A, the highest dose of LEO 138559 [Temtokibart], given every week from Week 0 to Week 3, then every 2 weeks from Week 4 to Week 16.
  LEO 138559: LEO 138559 [Temtokibart] given by injection just under the skin
- Dose Regimen 2: Dose B, medium-high dose of LEO 138559 [Temtokibart], given every week from Week 0 to Week 2, then every 2 weeks from Week 4 to Week 16.
  LEO 138559: LEO 138559 [Temtokibart] given by injection just under the skin
- Dose Regimen 3: Dose A, highest dose of LEO 138559 [Temtokibart], given at Week 0 and Week 2, then dose C (medium-low dose of LEO 138559 [Temtokibart]) every 2 weeks from Week 4 to Week 16.
  LEO 138559: LEO 138559 [Temtokibart] given by injection just under the skin
- Dose Regimen 4: Dose C, medium-low dose of LEO 138559 [Temtokibart], given at Week 0 and Week 2, then dose D (lowest dose of LEO 138559 [Temtokibart]) every 2 weeks from Week 4 to Week 16
  LEO 138559: LEO 138559 [Temtokibart] given by injection just under the skin
- Placebo Regimen: Placebo every week from Week 0 to Week 3, then every 2 weeks from Week 4 to Week 16
  Placebo: Placebo given by injection just under the skin. Placebo contains no active ingredients.
Period: Overall Study
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Placebo Regimen
Started | 52 | 53 | 52 | 53 | 52
Completed | 40 | 45 | 40 | 38 | 35
Not Completed | 12 | 8 | 12 | 15 | 17
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 1
Not completed — Lack of Efficacy | 1 | 2 | 1 | 1 | 6
Not completed — Withdrawal by Subject | 8 | 4 | 8 | 10 | 8
Not completed — Lost to Follow-up | 2 | 1 | 1 | 1 | 1
Not completed — Protocol-specified withdrawal criteria, withdrawal by investigator, prohibited medication used | 1 | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo Regimen: Placebo every week from Week 0 to Week 3, then every 2 weeks from Week 4 to Week 16.
  Placebo: Placebo given by injection just under the skin. Placebo contains no active ingredients.
- Total: Total of all reporting groups
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Placebo Regimen | Total
Number analyzed (Participants) | 52 | 53 | 52 | 53 | 52 | 262
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (13.8) | 35.7 (14.3) | 39.0 (15.7) | 35.9 (14.4) | 32.1 (11.1) | 35.5 (14.0)
Age, Customized [Count of Participants; unit: Participants]
  18 to <65 years | 50 | 51 | 50 | 50 | 52 | 253
  65 to <85 years | 2 | 2 | 2 | 3 | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 24 | 26 | 28 | 26 | 130
  Male | 26 | 29 | 26 | 25 | 26 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7 | 4 | 2 | 20
  Not Hispanic or Latino | 42 | 42 | 41 | 47 | 44 | 216
  Unknown or Not Reported | 7 | 7 | 4 | 2 | 6 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 12 | 9 | 13 | 11 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 5 | 0 | 2 | 3 | 0 | 10
  White | 33 | 34 | 36 | 35 | 34 | 172
  More than one race | 0 | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 7 | 6 | 4 | 2 | 6 | 25
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 4 | 7 | 4 | 3 | 20
  Romania | 1 | 1 | 0 | 0 | 0 | 2
  Hungary | 1 | 0 | 2 | 3 | 2 | 8
  United States | 6 | 3 | 5 | 8 | 4 | 26
  Czechia | 5 | 5 | 4 | 5 | 6 | 25
  Japan | 6 | 7 | 7 | 7 | 7 | 34
  Poland | 12 | 9 | 9 | 11 | 13 | 54
  United Kingdom | 2 | 2 | 3 | 2 | 5 | 14
  France | 7 | 5 | 4 | 1 | 6 | 23
  Germany | 7 | 13 | 7 | 7 | 4 | 38
  Spain | 3 | 4 | 4 | 5 | 2 | 18
EASI score [Mean (Standard Deviation); unit: scores on a scale] — The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe, and/or more extensive condition.
  scores on a scale | 25.74 (9.51) | 25.61 (8.95) | 26.73 (11.28) | 26.53 (10.41) | 26.13 (10.97) | 26.15 (10.19)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Eczema Area and Severity Index (EASI) Score
Description: The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of atopic dermatitis. The EASI is a composite index with scores ranging from 0 to 72, with higher values indicating more severe, and/or more extensive condition.
Time Frame: From baseline to Week 16
Population: For the primary efficacy endpoint, analyzed population was Full Analysis Set (FAS).
Measure: Least Squares Mean (95% Confidence Interval); unit: percent of change
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Placebo Regimen
Number analyzed (Participants) | 52 | 53 | 52 | 53 | 52
percent of change | -61.15 [-71.38 to -50.91] | -57.05 [-67.13 to -46.96] | -64.27 [-74.55 to -53.99] | -51.42 [-61.91 to -40.92] | -41.74 [-52.18 to -31.31]
Statistical Analysis 1: Comparison: Dose Regimen 1 vs Placebo Regimen; Study uses a hierarchical testing procedure to control the familywise error rate at 5% significance level. Null hypotheses are tested sequentially according to decreasing dose. Sequential testing procedure continues if the null hypothesis is rejected. For the primary estimand for the primary endpoint, initiation of rescue treatment and permanent discontinuation of IMP are considered intercurrent events; Test type: Superiority — Data following rescue treatment and permanent IMP discontinuations due to lack of effect or an AE related to worsening of AD will be considered missing not at random and imputed using LOCF. Data following other intercurrent events will also be set to missing, and will, together with other naturally occurring missing data, be imputed from a linear model assuming missing at random; p = 0.0090, ANCOVA — Imputed datasets are analyzed using ANCOVA model adjusted for treatment, baseline vIGA-AD score, baseline value, region, prior use of biologics or systemic JAKis for AD. Estimates are combined across the imputed datasets using Rubin's rule; Mean Difference (Net) = -19.40, 95% CI 2-sided [-33.96 to -4.84]
Statistical Analysis 2: Comparison: Dose Regimen 2 vs Placebo Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0393, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -15.3, 95% CI 2-sided [-29.85 to -0.75]
Statistical Analysis 3: Comparison: Dose Regimen 3 vs Placebo Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0026, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -22.52, 95% CI 2-sided [-37.18 to -7.87]
Statistical Analysis 4: Comparison: Dose Regimen 4 vs Placebo Regimen; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.1993, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Net) = -9.67, 95% CI 2-sided [-24.44 to 5.10]

2. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: An event will be considered treatment emergent if started after the first dose of IMP or if started before the first dose of IMP and worsened in severity after first dose of IMP.
Time Frame: From baseline (Week 0) to Week 16
Population: For the safety analysis, analyzed population was Safety Analysis Set (SAF).
Measure: Number; unit: adverse events
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Placebo Regimen
Number analyzed (Participants) | 52 | 53 | 52 | 53 | 52
adverse events | 98 | 124 | 83 | 118 | 78

ADVERSE EVENTS:
Time Frame: 32 weeks (Treatment period: Week 0 to Week 16; Safety follow-up period: Week 16 to Week 32)
Description: An event will be considered treatment emergent if started after the first dose of IMP or if started before the first dose of IMP and worsened in severity after first dose of IMP. An event will not be considered treatment-emergent if starting 18 weeks after the last dose of IMP. Any event that occurred prior to IMP administration was not considered treatment-emergent, as it was not triggered by the intervention.
Groups:
- Placebo Regimen: Placebo every week from Week 0 to Week 3, then every 2 weeks from Week 4 to Week 16 Placebo: Placebo given by injection just under the skin
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Placebo Regimen
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/53 | 0/52 | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 1/52 | 2/53 | 1/52 | 2/53 | 0/52
Other Adverse Events (participants affected / at risk) | 27/52 | 27/53 | 24/52 | 31/53 | 21/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Regimen 1 (N=52) | Dose Regimen 2 (N=53) | Dose Regimen 3 (N=52) | Dose Regimen 4 (N=53) | Placebo Regimen (N=52)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Regimen 1 (N=52) | Dose Regimen 2 (N=53) | Dose Regimen 3 (N=52) | Dose Regimen 4 (N=53) | Placebo Regimen (N=52)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 6 (6) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 5 (5) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 15 (18) | 11 (15) | 9 (13) | 13 (15) | 11 (13)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (6) | 3 (5) | 2 (2) | 1 (1) | 2 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (6) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 4 (4) | 10 (12) | 12 (17) | 15 (24) | 12 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
LEO Pharma seeks publication of all Phase 3 clinical trials in peer-reviewed journals within 12 months of trial completion, regardless of whether the findings are positive or negative. If there is no multi-centre publication within 12 months after the clinical trial has been completed or terminated at all trial sites, the investigator has the right to publish the results from the clinical trial generated by the investigator.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT05923099/Prot_SAP_000.pdf